CLINICAL TRIAL: NCT05034354
Title: Development and Feasibility of a Virtual Remote Physiological Monitoring Program of Children With Heart Disease
Brief Title: Virtual Remote Physiological Monitoring Program of Children With Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00112366
Record Dates: First submitted 2021-08-27; First posted 2021-09-05 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Pediatric ALL; Congenital Heart Disease; Single-ventricle; Biventricular Congestive Heart Failure; Heart Failure; Heart Failure，Congestive; Transplant; Failure, Heart
Keywords: Remote physiological monitoring; Qualitative interviews; Perceptions of virtual care
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Heart Defects, Congenital; Univentricular Heart; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective multi-methods observational study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote physiological monitoring (Experimental): Patients will be recruited from inpatient and outpatient cardiology service at the Stollery Children's Hospital will be purposively selected, with 50% of the patients living at least 100km from the Stollery into one of the following groups:
  Group 1: Infants <12 months of age with single ventricle physiology or biventricular cyanotic congenital heart disease.
  Group 2: Patients aged 5-17 with heart failure, listed for transplant, or within 1 year of transplant.
  Interventions: Device: Remote physiological monitoring

INTERVENTIONS:
Device: Remote physiological monitoring — Participants will be provided with a Bluetooth capable weight scale (A&D Medical UC-352BLE or Beurer BY90), oxygen saturation monitor (Contec Medical Systems CMS50D-BT) and automatic blood pressure monitor (A&D Medical UA- 651BLE) to use daily for at least 10 days of a 14-day trial period. Data will be sent via the Sphygmo App to the pediatric cardiology for monitoring. Parents and healthcare providers will be asked to participate in a qualitative interview and the end of the 14-day period to provide feedback on the devices and Sphygmo™ platform.

SUMMARY:
Infants and children with heart conditions require treatment in children's hospitals that are typically located in large cities. This creates challenges for children and families who need to travel long distances to come to appointments. Providing quality care to children with heart disease has further been challenged by the COVID-19 pandemic, with a shift towards decreased in-person contact and an increase in virtual visits, where assessment by doctors and nurses is more limited.

This research study will look at how families of children with heart disease access care and how investigators can improve care with virtual technologies. This will involve testing a new home-based virtual care platform that uses Bluetooth technology to connect weight scales, oxygen measuring devices and blood pressure cuffs with a smartphone app, allowing parents to easily use these devices and send accurate data directly to the cardiology team. Investigators will obtain feedback from families, patients, and healthcare providers about how this helped or did not help them, and adjust the technology as needed to make it better.

DETAILED DESCRIPTION:
This will be a prospective multi-methods observational study. Investigators will assess the feasibility of the novel home-based remote physiological monitoring (RPM) system paired to a smartphone app (Sphygmo™) and linked to a secure physician platform. The study team will enroll caregivers of medically high- risk infants with CHD and children and caregivers with heart failure or early post heart transplant. In addition, investigators will obtain feedback from their healthcare providers. Qualitative analysis of semi- structured interviews will determine patient and parent/caregiver and healthcare providers experience with the system and allow for future modifications specific to pediatrics.

Purposive sampling will be used to achieve a maximum variation and will ensure a diverse group of patients/caregivers that represent a variety of patient profiles. The study team aim to recruit 10 participants in each group, with 50% of the patients living at least 100 km drive from the Stollery.

Medical records will be accessed to collect baseline characteristics including date of birth, sex, postal code, diagnoses, surgeries and procedures. The number of pediatric cardiology clinic visits, hospitalizations, ED visits, and cardiac investigations in the last 2 years will be collected to describe the patients requirements for access to cardiac care. In addition, the family will be asked to complete a demographic form that compiles information about parents' ethnicity, education level, SES, access to Wi-FI and iOS/Android devices in the home.

An emerging, qualitative descriptive approach will be used to explore patient and parents' experiences using the RPM devices and app in their home as part of their daily care routine. Data collection and analysis will occur iteratively to allow emerging ideas. Semi-structured interviews with parents/patients/healthcare providers will be conducted by a qualitatively trained members of the study team. Data collection will occur until saturation (data redundancy) is achieved. Interviews will be held and recorded on a secure, password protected Zoom™ ECHO account and digitally captured and transcribed by Zoom auto-transcription services.

Baseline and demographic characteristics will be analyzed using descriptive statistics. Investigators will ascertain adherence with the protocol by determining the mean number of requested assessments performed and the proportion of patients who completed >80% of measurements. This will contribute to our understanding of the acceptability of this technology from the patient and family perspective.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Pediatric Cardiology at the Stollery Children's Hospital in Edmonton, AB
* Group 1: infants <12 months of age with single ventricle physiology or biventricular cyanotic congenital heart disease
* Group 2: patients aged 5 to 17 years with heart failure, listed for heart transplant, or within 1-year of heart transplant
* English speaking
* Access to internet either in the household or within the community

Exclusion Criteria:

* Inability to use technology due to physical or cognitive impairment in the caregiver
* Non-English speaking (thus limiting communication during qualitative interviews)
* No access to the internet (thus unable to transmit the device data through the app or be able to complete the qualitative interview)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Acceptability of technology | 3-weeks
  We will ascertain adherence with the protocol by determining the mean number of requested assessments performed and the proportion of participants who complete >80% of measurements. This will contribute to our understanding of the acceptability of this technology from the patient and family perspective.

SECONDARY OUTCOMES:
Device and app feedback | 3-weeks
  Families, participants if they are of age and understanding, and healthcare providers will provide feedback through qualitative interviews on the Bluetooth devices and Sphygmo application. As the app is designed for adults, this feedback will allow the study team to work with developers on a pediatric focused version of the application.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Conway, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorch SA, Rogowski J, Profit J, Phibbs CS. Access to risk-appropriate hospital care and disparities in neonatal outcomes in racial/ethnic groups and rural-urban populations. Semin Perinatol. 2021 Jun;45(4):151409. doi: 10.1016/j.semperi.2021.151409. Epub 2021 Mar 21. PMID 33931237
- [Background] Choi SA, Lim K, Baek H, Yoo S, Cho A, Kim H, Hwang H, Kim KJ. Impact of mobile health application on data collection and self-management of epilepsy. Epilepsy Behav. 2021 Jun;119:107982. doi: 10.1016/j.yebeh.2021.107982. Epub 2021 May 1. PMID 33946011
- [Background] Padwal R, Wood PW. Digital Health Approaches for the Assessment and Optimisation of Hypertension Care Provision. Can J Cardiol. 2021 May;37(5):711-721. doi: 10.1016/j.cjca.2020.12.009. Epub 2020 Dec 17. PMID 33340672
- [Background] Padwal RS, So H, Wood PW, Mcalister FA, Siddiqui M, Norris CM, Jeerakathil T, Stone J, Valaire S, Mann B, Boulanger P, Klarenbach SW. Cost-effectiveness of home blood pressure telemonitoring and case management in the secondary prevention of cerebrovascular disease in Canada. J Clin Hypertens (Greenwich). 2019 Feb;21(2):159-168. doi: 10.1111/jch.13459. Epub 2018 Dec 20. PMID 30570200
- [Background] Hehir DA, Ghanayem NS. Single-ventricle infant home monitoring programs: outcomes and impact. Curr Opin Cardiol. 2013 Mar;28(2):97-102. doi: 10.1097/HCO.0b013e32835dceaf. PMID 23337893
- [Background] Siehr SL, Norris JK, Bushnell JA, Ramamoorthy C, Reddy VM, Hanley FL, Wright GE. Home monitoring program reduces interstage mortality after the modified Norwood procedure. J Thorac Cardiovasc Surg. 2014 Feb;147(2):718-23.e1. doi: 10.1016/j.jtcvs.2013.04.006. Epub 2013 May 8. PMID 23663957
- [Background] Castellanos DA, Herrington C, Adler S, Haas K, Ram Kumar S, Kung GC. Home Monitoring Program Reduces Mortality in High-Risk Sociodemographic Single-Ventricle Patients. Pediatr Cardiol. 2016 Dec;37(8):1575-1580. doi: 10.1007/s00246-016-1472-x. Epub 2016 Aug 23. PMID 27554255
- [Background] Park KT, Bensen R, Lu B, Nanda P, Esquivel C, Cox K. Geographical rural status and health outcomes in pediatric liver transplantation: an analysis of 6 years of national United Network of Organ Sharing Data. J Pediatr. 2013 Feb;162(2):313-8.e1. doi: 10.1016/j.jpeds.2012.07.015. Epub 2012 Aug 20. PMID 22914224
- [Background] Bertagnin E, Greco A, Bottaro G, Zappulla P, Romanazzi I, Russo MD, Lo Presti M, Valenti N, Sollano G, Calvi V. Remote monitoring for heart failure management during COVID-19 pandemic. Int J Cardiol Heart Vasc. 2021 Feb;32:100724. doi: 10.1016/j.ijcha.2021.100724. Epub 2021 Jan 28. PMID 33532544